CLINICAL TRIAL: NCT05814341
Title: The Effect of Increasing Post-Filter Ionized Target on the Efficacy of Regional Citrate Anticoagulation During Continuous Renal Replacement Therapy in Intensive Care: a Multicenter Randomized Controlled Non-Inferiority Trial
Brief Title: Citrate Anticoagulation in Renal Replacement Therapy: Impact of a High Post-filter Calcium Target on Efficacy
Acronym: Ca-CIBLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220257; 2022-003678-22 (Other: ANSM)
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-07

CONDITIONS: Renal Replacement Therapy
Keywords: Acute kidney injury; Continuous renal replacement therapy; Regional citrate anticoagulation; Ionized calcium; Intensive care
MeSH Terms: conditions — Acute Kidney Injury | interventions — Citric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High iCa target (Experimental): Post-filter iCa between 0,35-0.45 mmol/L
  Interventions: Drug: Citrate
- Low iCa target (Active Comparator): Post-filter iCa between 0.25-0.35 mmol/L
  Interventions: Drug: Citrate

INTERVENTIONS:
Drug: Citrate — Comparison of two dosage adjustment protocols for medication according to different post-filter iCa targets
  Other Names: REGIOCIT®

SUMMARY:
Regional citrate anticoagulation (RCA) is the recommended method for anticoagulation in continuous renal replacement therapy (CRRT). However, the optimal post-filter ionized calcium (iCa) target level remains unclear. Currently, it is titrated to a post-filter iCa target ranging from 0.25 to 0.35 mmol/L, which is derived from a few underpowered trials. There are potential side effects associated with citrate administration, which may be increased in patient with liver failure and/or tissue dysoxia, such as alkalemia, acidemia, hypernatremia, hypocalcemia, hypomagnesemia, and citrate accumulation. Consequently, citrate anticoagulation is contraindicated in the most severe cases. The challenge is to use the minimum necessary dose of citrate to ensure both effective anticoagulation of the circuit and limit citrate administration to reduce the risks of metabolic complications and accumulation. This approach expands the indications for citrate, standardizes practice, and reduces financial costs. Investigators hypothesized that increasing the post-filter iCa target in RCA can limit the dose of citrate, thereby avoiding adverse effects (safety) without compromising the effectiveness of the treatment in preventing filter clotting. The aim of this study is to evaluate the impact of an increased post-filter iCa target from 0.25-0.35 to 0.35-0.45 mmol/L on the incidence of filter clotting for RCA-CRRT in critically ill patients. Investigators are designing a multicenter randomized controlled non-inferiority study.

DETAILED DESCRIPTION:
RCA-CRRT will be ordered based on clinical indications and will be performed according to a standardized protocol (available as online supplementary material) in continuous veno-venous hemofiltration mode with the same system (Prismaflex®; Gambro-Baxter, Deerfield, IL, USA) and a 0.9 m2 high-flux AN69 membrane. Blood flow will be maintained between 120 and 180 mL/min according to the patient's ideal body weight. The prescribed dose of filtration will be 30 mL/kg/h to achieve a delivered dose of 20-25 mL/kg/h, following KDIGO guidelines. A citrated replacement solution (Regiocit®; Gambro-Baxter), containing 18.0 mmol/L of citrate, will be delivered continuously to the blood before the filter of the extracorporeal circuit. The rate of infusion of predilution replacement flow will be coupled to the blood flow, aiming for a stable citrate concentration in the extracorporeal circuit. The initial citrate dose will be 3.0 mmol/L of blood, and then citrate flow rate will be adjusted to the post-filter iCa target according to the protocol. Post-filter iCa will be measured on ABL90 FLEX PLUS™ (Radiometer Medical©, Copenhagen, Denmark) blood gas analyzer 15 minutes after any change in dose and then every 6 hours. Calcium chloride will be administered to the patient through a central line to maintain systemic-iCa within 1.00-1.30 mmol/L. Fluid removal rates will be left to the discretion of the attending physician in order to achieve optimal fluid balance. Additionally, metabolic monitoring will be carried out by a blood ionogram every 12 hours. The quantitative parameters will be presented as median and interquartile range [IQR], and comparisons will be made using either Student's t-test or the Mann-Whitney U test depending on whether the assumptions of the t-test are met or not. Categorical data will be reported as the number and percentage (%) and will be compared using Fisher's exact or chi-square test, as appropriate. The incidence of filter clotting will be expressed in absolute values (n) and percentage (%). Comparison between groups will be performed using Pearson's Chi-square test. The analysis of the primary endpoint will be conducted on a per-protocol basis as a first intention (the most conservative approach in a non-inferiority study) and on an intention-to-treat basis. Filter lifespan until clotting curves according to the post-filter iCa2 target will be plotted using the Kaplan-Meier method and compared using the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Hospitalized in intensive care and presenting an indication for extra renal replacement therapy with Regional citrate anticoagulation (RCA)
3. Patients covered by social security regimen (excepting AME)
4. Having given their written consent or, if the patient is unable to consent and is accompanied, written consent from or legal representative or the close relative. If the patient is unable to consent and is not accompanied, due to the urgency of the procedure, the patient can also be included on the decision of the investigator (inclusion procedure in an emergency situation with subsequent necessity to sign a consent to prosecute).

Exclusion Criteria:

1. Patients receiving curative systemic anticoagulation
2. Patients with a contraindication to the use of citrate : - Hypersensitivity to Regiocit®
3. Patients with a contraindication to the administration of the ancillary drugs Phoxilium® and calcium chloride
4. Patients with an absolute contraindication to the use of citrate due to a lack of metabolism in the Krebs cycle and therefore a major risk of accumulation:

   * Severe impairment of liver function with PT < 30% and lactates > 3mmol/l
   * Severe tissue dysoxia in uncontrolled shock with lactic acidosis (lactates > 4mmol/l)
   * Drug toxicity (metformin, paracetamol, propofol, cyclosporine)
5. Pregnant woman
6. People under legal protection measure (guardianship or safeguard measures)
7. A patient legal representative or the close relative who declined to participate
8. Patient deprived of liberty by a judicial or administrative decision
9. Patient participating to another interventional study that may have an impact on the evaluation criteria of this study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of filter clotting | 72 hours
  Filter clotting was defined by increased transmembrane pressure greater than 300 mmHg
Incidence of filter clotting | 72 hours
  Filter clotting was defined by visible thrombus in circuit or filter
Incidence of filter clotting | 72 hours
  Filter clotting was defined by inability to rotate the blood pump due to an obstructing thrombus

SECONDARY OUTCOMES:
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by filter clotting
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by catheter dysfunction : excessively negative inlet pressure (less than -150mmHg) or excessively positive outlet pressure (greater than +150mmHg)
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by transport: removal of the patient for mobilization
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by futility: no indication to continue CRRT
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by end of session: CRRT has been ongoing for more than 72 hours
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by citrate accumulation
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by Intensive Care Unit discharge
Filter lifespan until clotting and filter lifespan, including all causes of stoppage | 72 hours
  The lifespan of each hemofilter measured in hours. The cause of CRRT discontinuation will be defined by death
Proportion of post-filter iCa in the target range and last psot-filter iCa value before clotting | 72 hours
  Post-filter iCa levels (in mmol/L) measured during the CRRT session
Total dose of citrate infused | 72 hours
  Citrate infusion rates, in mmol/day
Incidence of metabolic events (hypocalcemia, metabolic acidosis, metabolic alkalosis, hypernatremia, hypomagnesemia, citrate accumulation) | 72 hours
  The occurrence of the following 6 metabolic complications:
  * Hypocalcemia [Ca2+ < 0.95mmol/L]
  * Metabolic acidosis [pH < 7.3 and HCO3- < 20mmol/L]
  * Metabolic alkalosis [pH > 7.5 and HCO3- > 30mmol/L]
  * Hypernatremia [Na+ > 145mmol/L]
  * Hypomagnesemia [Mg2+ < 0.70mmol/L]
  * Citrate accumulation [total calcium/ionized calcium ratio > 2.5]
Financial costs associated with filter changes and citrate use | 72 hours
  The costs (in euros) incurred by each filter change and the amount of citrate infused
Blood loss during the procedure | 72 hours
  Inability to return the CRRT circuit at the end of the session (equivalent to 200mL of blood loss)

CONTACTS AND LOCATIONS:
Overall Officials: Mona ASSEFI, Dr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hospital Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Derived] Assefi M, Braik R, James A, Clavieras N, Baron E, Blanchard F, Constantin JM. Impact of increasing post-filter ionised calcium target on regional citrate anticoagulation efficacy in ICU continuous renal replacement therapy: the non-inferiority randomised controlled Ca-CIBLE protocol. BMJ Open. 2024 Sep 26;14(9):e081325. doi: 10.1136/bmjopen-2023-081325. PMID 39327056